CLINICAL TRIAL: NCT03934814
Title: A Phase 1 Study of TJ011133 Administered Alone or in Combination With Pembrolizumab or Rituximab in Subjects With Relapsed/Refractory Advanced Solid Tumors and Lymphoma
Brief Title: Study of TJ011133 in Participants With Relapsed/Refractory Advanced Solid Tumors and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TJ011133EDI101; KEYNOTE A21 (Registry Identifier: Merck Sharp & Dohme LLC); MK-3475-A21 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor; Lymphoma
Keywords: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1A - TJ011133 Monotherapy (Experimental): TJ011133 alone will be administered at up to 7 dose levels (0.3, 1, 3, 10, 20, 30, 45 mg/kg) once weekly (Q1W) (the 0.3 mg/kg dose level cohort will be enrolled if a DLT in 1 out of 3 subjects is observed following the 1 mg/kg dose level).
  Interventions: Drug: TJ011133
- Part 1B - Combination therapy of TJ011133 with pembrolizumab (Experimental): TJ011133 will be administered Q1W, starting at 20 mg/ kg, in combination with pembrolizumab.
  Interventions: Drug: TJ011133; Drug: Pembrolizumab
- Part 1C - Combination therapy of TJ011133 with rituximab (Experimental): TJ011133 will be administered Q1W, starting at 20 mg/kg, in combination with rituximab.
  Interventions: Drug: TJ011133; Drug: Rituximab
- Part 2 - Dose Expansion (Experimental): 30 participants (with DLBCL or indolent lymphoma) in the TJ011133 combination therapy with rituximab expansion and 20 participants with solid tumors in the TJ011133 combination therapy with pembrolizumab expansion.
  Interventions: Drug: TJ011133; Drug: Pembrolizumab; Drug: Rituximab

INTERVENTIONS:
Drug: TJ011133 — TJ011133 will be administered weekly.
Drug: Pembrolizumab — Pembrolizumab will be administered every 3 weeks.
  Other Names: KEYTRUDA®
  Arms: Part 1B - Combination therapy of TJ011133 with pembrolizumab; Part 2 - Dose Expansion
Drug: Rituximab — Rituximab will be administered weekly for 5 doses, then followed by monthly doses.
  Other Names: Rituxan; MabThera
  Arms: Part 1C - Combination therapy of TJ011133 with rituximab; Part 2 - Dose Expansion

SUMMARY:
The purpose of this study is to assess the safety and tolerability of TJ011133 in participants with solid tumors and lymphoma.

DETAILED DESCRIPTION:
This is an open-label, multi-center, multiple dose, Phase 1 study to evaluate the safety, tolerability, maximum tolerated dose (MTD) or maximum administered dose (MAD), pharmacokinetic (PK), pharmacodynamic, and recommended Phase 2 dose (RP2D) of TJ011133, an anti-CD47 antibody, in participants with advanced relapsed or refractory solid tumors and lymphoma. The study will be conducted in 2 parts. Part 1 comprises a single agent dose escalation (Part 1A) and 2 separate combination therapy dose escalations (Part 1B with pembrolizumab and Part 1C with rituximab) and Part 2 includes a dose expansion study.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Participants with advanced relapsed/refractory solid tumors and lymphoma.
* Part 2 with Rituximab: Participants with diffuse large B-cell lymphoma (DLBCL) or Indolent B-cell Lymphoma, with at least one measurable lesion by Lugano and available fresh metastatic biopsy sample prior to study entry.
* Part 2 with Pembrolizumab: Participants with locally advanced non-small-cell lung carcinoma (NSCLC) with disease progression or immune-oncology treatment naive Epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer, with at least one measurable lesion defined by Response Elevation Criteria in Solid Tumors (RECIST) 1.1, and available fresh metastatic biopsy prior to study entry.
* All Parts: Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1 and adequate bone marrow, renal, and liver functions.

Exclusion Criteria:

* Participants with known symptomatic central nervous system tumors or known central nervous system metastases or leptomeningeal disease requiring steroids. Participants who document stable and central nervous system metastases and are off steroids for more than 4 weeks may be enrolled in the study.
* Participants with Burkitt's lymphoma, lymphoblastic lymphoma, Richter's transformation, primary effusion lymphoma or chronic lymphocytic leukemia/small lymphocytic lymphoma.
* Participants with mantle cell lymphoma.
* Impaired cardiac function or clinically significant cardiac diseases.
* Prior treatment with CD47 or SIRPα inhibitors.
* Prior autologous stem cell transplant <=3 months prior to starting study.
* Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning.
* Prior chimeric antigen receptor or chimeric antigen receptor T-cell therapy.
* History of autoimmune anemia or autoimmune thrombocytopenia.
* Positive Direct Antiglobulin Test.
* Active graft versus host disease (GVHD) or ongoing immunosuppression for GVHD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 21 or 28 days, depending on study part
  Part 1A DLT period is 3 weeks, Part 1B DLT period is 3 weeks, Part 1C DLT period is 4 weeks.
Incidence and Severity of Adverse Events | up to 100 days post last dose
  The CTCAE criteria will be used to assess adverse events on this trial.
Maximum Tolerated Dose (MTD) for Both Monotherapy and Combination Therapy | 21 or 28 days, depending on study part
  Based on DLT definitions.
Change in Eastern Cooperative Oncology Group (ECOG) Performance Status | up to 100 days post last dose
  Change in Eastern Cooperative Oncology Group (ECOG) Performance Status.

SECONDARY OUTCOMES:
Pharmacokinetic (PK): Area Under the Curve From Time Zero To Infinity (AUC∞) | up to 100 days post last dose
  Area under the curve from time zero to infinity (AUC∞).
PK: Area Under the Curve From Time Zero To The Time Of The Last Quantifiable Concentration (AUC0-t) | up to 100 days post last dose
  Area under the curve from time zero to the time of the last quantifiable concentration (AUC0-t).
PK: Maximum Observed Concentration (Cmax) | up to 100 days post last dose
  Maximum observed concentration (Cmax).
PK: Time of the Maximum Observed Concentration (Tmax) | up to 100 days post last dose
  Time of the maximum observed concentration (Tmax).
PK: Terminal Elimination Half-Life (T1/2) | up to 100 days post last dose
  Investigational Product (IP) terminal elimination half-life (T1/2).
PK: Clearance (CL) | up to 100 days post last dose
  Investigational Product (IP) Clearance (CL).
PK: Volume Of Distribution (Vz) | up to 100 days post last dose
  Investigational Product (IP) volume of distribution (Vz).
PK: AUC Over A Dosing Interval (AUCtau) | up to 100 days post last dose
  AUC over a dosing interval (AUCtau).
PK: Trough Concentration (Ctrough) | up to 100 days post last dose
  Investigational Product (IP) trough concentration (Ctrough).
PK: Volume of Distribution at Steady State (Vss) | up to 100 days post last dose
  Investigational Product (IP) volume of distribution at steady state (Vss).
Immunogenicity: Anti-drug antibodies (ADA) | up to 100 days post last dose
  Incidence and concentration of anti-drug antibodies.
Efficacy: Best Overall Response (BOR) | up to 100 days post last dose
  BOR is determined using Response Elevation Criteria in Solid Tumors (RECIST) 1.1 and immune Response Elevation Criteria in Solid Tumors (iRECIST) guidelines for response criteria for use in trials testing immunotherapeutics for solid tumors and Lugano criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma.
Efficacy: Objective Response Rate (ORR) | up to 100 days post last dose
  ORR is determined using Response Elevation Criteria in Solid Tumors (RECIST) 1.1 and immune Response Elevation Criteria in Solid Tumors (iRECIST) guidelines for response criteria for use in trials testing immunotherapeutics for solid tumors and Lugano criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma.
Efficacy: Duration Of Response (DOR) | up to 100 days post last dose
  DOR is determined using Response Elevation Criteria in Solid Tumors (RECIST) 1.1 and immune Response Elevation Criteria in Solid Tumors (iRECIST) guidelines for response criteria for use in trials testing immunotherapeutics for solid tumors and Lugano criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma.
Efficacy: Progression-Free Survival (PFS) | up to 100 days post last dose
  PFS is determined using Response Elevation Criteria in Solid Tumors (RECIST) 1.1 and immune Response Elevation Criteria in Solid Tumors (iRECIST) guidelines for response criteria for use in trials testing immunotherapeutics for solid tumors and Lugano criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma.
Efficacy: Overall Survival (OS) | up to 100 days post last dose
  OS is determined using Response Elevation Criteria in Solid Tumors (RECIST) 1.1 and immune Response Elevation Criteria in Solid Tumors (iRECIST) guidelines for response criteria for use in trials testing immunotherapeutics for solid tumors and Lugano criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Yale School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Horizon Oncology, Lafayette, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer Institute/Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Fourth Hpspital of Hebei Medical University(Hebei Cancer Hospital), Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - HuBei Cancer Hospital, Wuhan, Hubei
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No